CLINICAL TRIAL: NCT05490303
Title: Development of Guidance Algorithms for Acquisition of Echocardiographic Reference Views
Brief Title: HeartGuide: Preliminary Study
Acronym: HG-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: DESKi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/19; 2022-A01501-42 (Other: ID-RCB)
Record Dates: First submitted 2022-07-29; First posted 2022-08-05 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Disease
Keywords: Echocardiography; Guidance algorithm
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other): Patient with an echocardiography examination
  Interventions: Other: recording of the probe position

INTERVENTIONS:
Other: recording of the probe position — For each patient, a cardiac ultrasound acquisition will be performed with an optical tracking system (infrared) recording the probe's position in real time.

SUMMARY:
Echocardiography is the examination of choice for the study of cardiac pathologies. Interest of echocardiography for other medical specialties has already been demonstrated (intensive care in the case of hemodynamic failure - in intra and extra hospital emergency medicine for the initial assessment of chest pain or dyspnea).

The expansion of echocardiography'use has been catalyzed by miniaturization of echographic systems and decrease in their price. Recently, probes directly connected to a tablet or phone have been developed at a limited cost.

Therefore, it's possible to consider these ultrasound scanners as the new stethoscope that could be used by any health professional.

The last limit to this democratization is the training, especially for non-specialists (non-cardiologists).

DETAILED DESCRIPTION:
Since January 2019, echocardiography laboratory headed by Prof. Stéphane Lafitte and DESKi (start-up - Bordeaux) have been working on guiding non-experts through their cardiac ultrasound examination.

An algorithm indicating in real time if the view obtained corresponds to a reference view has already been validated. However, this algorithm does not tell the operator which movement would improve the image quality.

Thanks to advances in deep learning and by combining cardiac ultrasound acquisitions with systems that record the position of the probes in real time, it would be possible to develop an algorithm able to guide the operator's movements.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) older than 18 years,
* Patient having a scheduled cardiac ultrasound outside any emergency context,
* Patients who have not objected to participating in the research (at the latest on the day of inclusion and before any examination required by the research),
* Subjects affiliated or benefiting from a social security plan,
* Women of childbearing age who are using effective contraception.

Exclusion Criteria:

* Person under legal protection (legal protection, guardianship or curatorship),
* Person deprived of liberty by judicial or administrative decision,
* Person who is unable to give his/her non-opposition,
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Probe position | Day 0
  Difference between actual probe position and predicted position with guidance algorithm

SECONDARY OUTCOMES:
Percentage of matches between algorithm and expert | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane LAFITTE, MD,PhD, Study Director — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France